CLINICAL TRIAL: NCT00967941
Title: Vancomycin and Daptomycin Plus Cefazolin for Preoperative Vascular Surgery Prophylaxis
Status: Completed | Type: Observational
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Patrick Stone, MD, Patrick Stone, MD,, CAMC Health System
Other Study IDs: 06-11-1879
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: MRSA Infections
Keywords: Vascular Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ancef
- Vancomycin and Cefazolin
- Daptomycin and Cefazolin

SUMMARY:
This study prospectively selects the patients to examine the effectiveness of the investigators' current standard of prophylaxis prior to vascular surgery and to compare the effectiveness of vancomycin and daptomycin plus cefazolin in reducing infections in vascular surgical patients.

DETAILED DESCRIPTION:
According to Medqic.org (site for the Surgical Care Improvement Project) the current recommended drug of choice for prophylaxis prior to vascular surgery is Cefazolin (Ancef). The exception would be to allow the use of Vancomycin as an acceptable antibiotic for patients undergoing cardiac, vascular or orthopedic surgery due to the increasing risk of methicillin-resistantStaphylococcus aureus (MRSA). The significance of the study is to demonstrate that MRSA coverage is needed in vascular surgery with prosthetic graft placement in areas of the body that is at high risk for infection. By decreasing post surgical site and prosthetic infections, we could significantly reduce vascular surgery mortality and morbidity. Cost and amputation rates we feel could also be reduced. patients will be randomized in three groups such as cefazolin,vancomycin and cefazolin, daptomycin and cefazolin and then patients will be monitored per usual post-operative course (30 days and 90 days follow-up) with wound and incision evaluation. Outcome measures include hospital length of stay, the presence of a graft infection, skin infection at incision site, vascular procedure failure secondary to infection, cost, thirty day readmits, amputation, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years of age undergoing vascular surgery including carotid procedures and a vascular access procedure (Fistula or Graft).

Exclusion Criteria:

* Patients with an allergy to daptomycin or vancomycin.
* Patients with chronic wounds.
* Prior colonization of MRSA.
* Increased MRSA rate facility wide.
* Continuous inpatient stay >27 hrs prior to surgical procedure.
* Patients with active infection requiring antibiotics preoperatively.
* Patients with a history of MRSA colonization or infection, HIV, admission for >3 months in an acute care center or long-term care center, penicillin allergy or penicillin allergy and on dialysis.
* Dialysis patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older undergoing a vascular surgery and or vascular access (vascular fistula or vascular graft) procedure were eligible for enrollment in the study.
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stone, M.D., Principal Investigator — CAMC Medical Staff-with admitting privileges
Locations (1):
- Vascular Center of Excellence, Charleston, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment was done during the period August 2007 through June 2009 at vascular center.
Pre-assignment Details: 12 patients were excluded from study for being ineligible due to active infection, dialysis, allergy to penicillin,NO procedure, withdrew from surgery.
Groups:
- Ancef: Ancef (Antibiotic Prophylaxis) : Comparing the antibiotic treatment related to surgery
- Daptomycin and Cefazolin: Daptomycin and Cefazolin (Antibiotic Prophylaxis) : Comparing the antibiotic treatment related to surgery
- Vancomycin and Cefazolin: Vancomycin and Cefazolin (Antibiotic Prophylaxis) : Comparing the antibiotic treatment related to surgery
Period: Overall Study
Arm/Group | Ancef | Daptomycin and Cefazolin | Vancomycin and Cefazolin
Started | 67 | 54 | 60
Completed | 62 | 51 | 56
Not Completed | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ancef | Daptomycin and Cefazolin | Vancomycin and Cefazolin | Total
Number analyzed (Participants) | 67 | 54 | 60 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.37 (11.78) | 66.78 (11.81) | 64.36 (11.12) | 65.17 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 20 | 66
  Male | 41 | 34 | 40 | 115

OUTCOME MEASURES:

1. Primary Outcome: Overall Number of Participants With Methicillin-resistant Staphylococcus Aureus (MRSA) Infections.
Time Frame: 30 days post-operative
Population: Patients with MRSA infections.
Measure: Number; unit: participants
Arm/Group | Ancef | Daptomycin and Cefazolin | Vancomycin and Cefazolin
Number analyzed (Participants) | 62 | 51 | 56
participants | 2 | 0 | 4

2. Secondary Outcome: Overall Groin Procedures in Patients With and Without Any Infection.
Time Frame: 30 days post-operative
Population: Patients with groin procedures.
Measure: Number; unit: Participants
Groups:
- Total Patients With Infection: Total number of patients who have infections in the study.
- Patients Without Infection: Total number of patients who do not have any infections.
Arm/Group | Total Patients With Infection | Patients Without Infection
Number analyzed (Participants) | 17 | 152
Participants | 14 | 83

ADVERSE EVENTS:
Description: Adverse Events were not collected and assessed as a part of this protocol.
Groups:
- All Patients: The adverse event was counted for all patients instead of groups. Ideally no unexpected adverse events. All were known risks in vascular procedures.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
We did not have standardization of skin preparation. Additionally, we did not have a specific protocol for dressing use and time of dressing removal. We excluded high-risk patients for MRSA infection in our study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No